CLINICAL TRIAL: NCT01752400
Title: A Phase II Open-Label Trial of AUY922, an HSP90 Inhibitor, in Patients With ALK-Rearranged Advanced Non-Small Cell Lung Cancer and Acquired Resistance to Prior ALK Tyrosine Kinase Inhibition
Brief Title: AUY922 for Advanced ALK-positive NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Alice Shaw, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-458
Record Dates: First submitted 2012-12-07; First posted 2012-12-19 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Advanced
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AUY922 (Experimental): Via intravenous infusion on Days 1, 8 and 15 of each 21 day cycle (once per week). Infusion lasts approximately 60 minutes
  Interventions: Drug: AUY922

INTERVENTIONS:
Drug: AUY922

SUMMARY:
This research study is a Phase II clinical trial, which tests the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific cancer. "Investigational" means that the drug is being studied and that research doctors are trying to find out more about it-such as the safest dose to use, the side effects it may cause and if the drug is effective for treating your type of cancer. It also means that the FDA has not yet approved the drug for your type of cancer or for any use outside of research studies.

It has been found that some people with NSCLC have a change (mutation) in a certain gene called the ALK gene. This mutated gene helps cancer cells grow. There is a drug (crizotinib) that has been approved by the FDA for the treatment of people with NSCLC who have mutations in the ALK gene. Most people respond to crizotinib initially. Over time, however, patients may stop responding (become resistant) to crizotinib because of additional changes in the ALK gene that makes crizotinib ineffective.

AUY922 is an investigational drug that may stop cancer cells from growing abnormally. This drug has been used in other research studies. Information from those other research studies suggests that AUY922 may be effective in killing cancer cells that have become resistant to drugs like crizotinib. Only participants with changes in the ALK gene will be allowed to participate in this study.

The purpose of this study is to test the safety of AUY922 and determine how well AUY922 treats participants with advanced, ALK-positive NSCLC.

DETAILED DESCRIPTION:
If you agree to participate in this research study, you will be asked to undergo some screening tests or procedures to find out if you can be in the research study. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated. These test include a medical history, physical exam, performance status, assessment of tumor, EKG, echocardiogram or multigated acquisition scan, eye exam, blood draw, blood pregnancy test, urine tset and collection of a piece of stored tumor tissue. If these tests show you are eligible to participate in the research study, you will begin the study treatment. If you do not meet the eligibility criteria, you will not be able to participate in this research study.

Study treatment is given in 21 day cycles. AUY922 is given by IV (into a vein). This is called an infusion. You will receive an infusion of AUY922 jon days 1,8 and 15 of each cycle (once per week). The infusion will take about 60 minutes.

A schedule of clinic visits for the study is summarized below. At every visit, you should tell the study staff how you are feeling and whether your health has changed. you may have other lab tests done as part of the the care of your cancer in addition to those listed below.

Cycle 1, Day 1: physical examination, performance status, EKG, Blood draw and routine urine tests.

Cycle 1, Day 2: EKG

Cycle 1, Day 3: EKG

Cycle 1, Day 8: measurement of weight and vital signs, performance status, EKG, questions about side effects you may have and medications you are taking

Cycle 1, Day 15: physical exam, performance status, EKG, blood draw, questions about side effects you may have and medications you are taking.

Note that in Cycle 1 you will need to stay at (or return to) the clinic for the last EKG following the Day 1 AUY922 infusion, and come to the clinic on Days 2 and 3 for EKGs

Cycle 2 and beyond, Day 1: physical exam, performance status, EKG, blood draw, questions about side effects you may have and medications you are taking, routine urine test

Cycle 2 and beyond, Day 8: measurement of weight and vital signs, performance status, EKG, questions about side effects and medications

Cycle 2 and beyond, Day 15: physical exam, vital signs, performance status, EKG, blood draw, questions about side effects and medications

Additional EKGs may be done at any time if your study doctor thinks it is necessary. A blood test to measure the amount of cardiac enzymes in your blood may be done whenever abnormal findings such as heart rhythm changes are suspected or seen on the EKG. CT or MRI scans will be done to measure your disease about every 6 weeks. A blood pregnancy test, for women who can become pregnant, will be performed every 6 weeks or at any point in which pregnancy is suspected. A standard eye exam will be done on Cycle 3, Day 1. Additional eye exams will be done if you experience any eye-related symptoms, such as changes in vision.

Within 1 week after your last dose of the study drug AUY922, you will be asked to return to the clinic for an End of Treatment Visit. At this visit the following will be done: physical examination, performance status, ECG, ECHO or MUGA scan, blood draw, urine test, eye exam, questions about side effects you may have and medications you are taking.

You will be asked to return to the clinic about 3 weeks after the End of Treatment Visit (about 4 weeks after the last dose of AUY922) so we can follow-up on any side effects you may still be experiencing after stopping AUY922.

If you decide to stop study treatment for a reason other than progression of your disease, you will be asked to have follow-up CT scans or MRIs every 12 weeks to continue to monitor the status of your cancer. If your tumors get worse, you will not need to have any further CT scans (or MRIs) as part of the study.

If your disease does progress, we would like to contact you by telephone about every 3 months to check on your status. This will be done until after the last participant stops study treatment, or for as long as you allow us to contact you. Keeping in touch with you and checking on your condition helps us look at the long term effects of the research.

You can continue to receive AUY922 for as long as your cancer does not progress and you do not experience unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced NSCLC
* Tumor characterized by abnormalities in ALK
* Required to provide archival tissue in the form of 5 formalin fixed paraffin embedded sections
* Have acquired resistance to treatment with an ALK-TKI
* At least one measurable lesion as defined by RECIST criteria
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Pregnant or breastfeeding
* Discontinued ALK TKI more than four weeks prior to enrollment
* Unresolved diarrhea greater than or equal to CTCAE grade 1
* Not willing to use double barrier methods of contraception
* Prior anti-neoplastic treatment with any HSP90 or HDAC inhibitor compound
* Have received cytoxic chemotherapy in the intervening period since discontinuation of an ALK-TKI
* Have undergone major surgery within 2 weeks prior to starting study drug
* Any concurrent or uncontrolled illness
* Any known disorders due to a deficiency in bilirubin glucuronidation
* Taking therapeutic doses of warfarin
* Any serious cardiac disorders or abnormalities
* Concurrent malignancies or invasive cancers diagnosed within the past 2 years except for adequately treated basal cell cancer of the skin or in situ cancers
* Known to be HIV positive
* Known hypersensitivity to any of the study drugs or their excipients
* Participation in another clinical study within 30 days before the first study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-01; Primary Completion 2017-06 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Shaw, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- AUY922: Via intravenous infusion on Days 1, 8 and 15 of each 21 day cycle (once per week). Infusion lasts approximately 60 minutes
  AUY922
Period: Overall Study
Arm/Group | AUY922
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AUY922
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 52.5 [42 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6
Region of Enrollment [Number; unit: participants]
  United States | 6
Smoking Status [Count of Participants; unit: Participants] — A pack year is the number of packs of cigarettes (1 pack= 20 cigarettes) smoked per day multiplied by the number of years smoking.
  Participants
    Never Smoker | 2
    Light Smoker (≤ 10 pack years) | 2
    Heavy Smoker (>10 pack years) | 2
Median Number of Prior Lines of Therapy [Median (Full Range); unit: Prior Lines of Therapy] | 3 [2 to 4]
Previous ALK Inhibitors [Number; unit: participants] — ALK: anaplastic lymphoma kinase
  Participants that received more than one ALK inhibitor were counted once for each inhibitor received
  participants
    Crizotinib | 5
    Alectinib | 1
    Certinib | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The number of participants that achieved either a complete response (CR) or a partial response (PR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to < 10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Baseline and then every six weeks (± 7 days), until the time of disease progression
Measure: Count of Participants; unit: Participants
Arm/Group | AUY922
Number analyzed (Participants) | 6
Participants | 0

2. Secondary Outcome: Progression-free Survival
Description: Progression free survival is measured as the number of months from date of study entry to date of progression or death, whichever comes first. Progression is assessed using RECIST v1.1.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study with at least a 5 mm absolute increase in the sum of all lesions. The appearance of one or more new lesions denotes disease progression.
Time Frame: From the start of treatment until the time of death or progression
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AUY922
Number analyzed (Participants) | 6
Months | 1.43 [1.3 to 2.8]

3. Secondary Outcome: Disease Control Rate
Description: The number of participants that achieved disease control, which includes complete responses, partial responses or stable disease as assessed by RECIST v1.1
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to < 10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Baseline and then every six weeks (± 7 days), until the time of disease progression
Measure: Count of Participants; unit: Participants
Arm/Group | AUY922
Number analyzed (Participants) | 6
Participants
  CR | 0
  PR | 3
  SD | 3

4. Secondary Outcome: Number of Participants Who Develop Adverse Events on AUY922
Description: The number of participants that developed any grade adverse event as assessed by Common Terminology Criteria for Adverse Events (CTCAE v4)
Time Frame: From the start of treatment until 30 days after last dose was received
Measure: Count of Participants; unit: Participants
Arm/Group | AUY922
Number analyzed (Participants) | 6
Participants | 6

5. Secondary Outcome: Number of Participants With Concurrent KRAS Mutations
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | AUY922
Number analyzed (Participants) | 6
Participants
  KRAS Mutation | 0
  Negative for KRAS Mutation | 2
  Unknown Mutation Status | 4

6. Secondary Outcome: ALK Translocation Variant Type
Time Frame: Baseline
Population: Data unavailable for all six participants
Arm/Group | AUY922
Number analyzed (Participants) | 0

7. Secondary Outcome: ALK Mutation Status
Description: The number of secondary ALK mutations or ALK amplification as a mechanism of resistance in pre-treatment and post-treatment biopsies.
Time Frame: Baseline, end of treatment
Population: Data not available for the other 5 participants
Measure: Count of Participants; unit: Participants
Arm/Group | AUY922
Number analyzed (Participants) | 1
Participants
  ALK Mutation | 1
  No ALK Mutation | 0

8. Secondary Outcome: Median Overall Survival
Description: The median duration of time from the start of treatment until the time of death or until the participant withdraws participation in the trial.
Time Frame: From the start of treatment until death or withdrawal from the study
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AUY922
Number analyzed (Participants) | 6
Months | 26.87 [9.03 to 26.87]

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after the last dose of the study drug was received. Treatment is continued until disease progression, unacceptable toxicity, participant withdrawal, death, or discontinuation from the study for any other reason.
Arm/Group | AUY922
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AUY922 (N=6)
Abdominal Pain (Gastrointestinal disorders) | 1 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AUY922 (N=6)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (2)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 4 (5)
Fatigue (General disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
INR increased (Investigations) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1)
Lung infection (Infections and infestations) | 1 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT01752400/Prot_SAP_000.pdf